CLINICAL TRIAL: NCT01202201
Title: A Retrospective Survey of the Burden of Rotavirus Gastroenteritis (RV GE) and Nosocomial RV GE in Children <6 Years of Age in Japan
Brief Title: A Retrospective Survey of the Burden of Rotavirus Gastroenteritis (RV GE) and Nosocomial RV GE in Japan
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114131
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Nosocomial Rotavirus Gastroenteritis; Rotavirus Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Study Cohort: Subjects hospitalized with acute gastroenteritis or rotavirus gastroenteritis
  Interventions: Other: Database analysis

INTERVENTIONS:
Other: Database analysis — Review and collect data from database (electronic admission database or any other applicable database of the hospital)

SUMMARY:
The purpose of this study is to evaluate the epidemiology and baseline disease burden of rotavirus gastroenteritis in children < 6 years of age, in Japan.

DETAILED DESCRIPTION:
This is a retrospective database study wherein data on children who have been diagnosed with acute gastroenteritis or rotavirus gastroenteritis will be collected from the electronic admission database or any other applicable database of the participating hospitals.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child aged <6 years at the time of admission in hospital. A child will become ineligible on the day of her/his sixth birthday.
* A subject who is hospitalized with any acute gastroenteritis or rotavirus gastroenteritis during the survey period.

Exclusion Criteria:

* Participants of any kind of rotavirus vaccine clinical trial.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children <6 years of age hospitalized with acute gastroenteritis or rotavirus gastroenteritis in any of the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 13767 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of acute gastroenteritis among all hospitalized children aged <6 years | At least 24 months (from 01 January 2008 to 31 December 2009)
Occurrence of rotavirus gastroenteritis among all hospitalized children aged <6 years | At least 24 months (from 01 January 2008 to 31 December 2009)
Occurrence of rotavirus gastroenteritis among all acute gastroenteritis hospitalizations in children aged <6 years | At least 24 months (from 01 January 2008 to 31 December 2009)

SECONDARY OUTCOMES:
Occurrence of nosocomial rotavirus gastroenteritis among all hospitalized children aged <6 years | At least 24 months (from 01 January 2008 to 31 December 2009)
Occurrence of nosocomial rotavirus gastroenteritis among all hospitalizations with rotavirus gastroenteritis in children aged <6 years | At least 24 months (from 01 January 2008 to 31 December 2009)
Prolongation of hospitalization of patients with nosocomial rotavirus gastroenteritis | At least 24 months (from 01 January 2008 to 31 December 2009)
Occurrence of rotavirus gastroenteritis hospitalization and nosocomial rotavirus gastroenteritis hospitalization among children <6 years of age, stratified by age | At least 24 months (from 01 January 2008 to 31 December 2009)
Seasonal distribution (monthly) of rotavirus gastroenteritis infection | At least 24 months (from 01 January 2008 to 31 December 2009)
Age (monthly) specific data of all the outcome measures, for children <12 months of age | At least 24 months (from 01 January 2008 to 31 December 2009)
Number of hospitalizations with rotavirus gastroenteritis and other vaccine-preventable infectious diseases such as influenza, mumps and varicella among children <6 years of age | At least 24 months (from 01 January 2008 to 31 December 2009)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Tajiri H, Takeuchi Y, Takano T, Ohura T, Inui A, Yamamoto K, Higashidate Y, Kawashima H, Toyoda S, Ushijima K, Ramakrishnan G, Rosenlund M, Holl K. The burden of rotavirus gastroenteritis and hospital-acquired rotavirus gastroenteritis among children aged less than 6 years in Japan: a retrospective, multicenter epidemiological survey. BMC Pediatr. 2013 May 22;13:83. doi: 10.1186/1471-2431-13-83. PMID 23697664